CLINICAL TRIAL: NCT04073771
Title: A Multiple Centre, Cohort Study of New Continuous Renal Replacement Therapy (CRRT) Membranes oXiris for Patients With Septic Shock
Brief Title: A Multiple Centre, Cohort Study of New CRRT Membranes oXiris for Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Songqiao Liu, Prof., Southeast University, China
Other Study IDs: 2018ZDSYLL152-P01; 18CECACAP1004 (Other Grant/Funding Number: Zhongda Hospital, Southeast University,)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Acute Kidney Injury Due to Sepsis (Disorder)
Keywords: Septic shock, AKI, CRRT
MeSH Terms: conditions — Shock, Septic | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort study: Patients with septic shock undergoing continuous renal replacement therapy
  Interventions: Device: Continuous renal replacement therapy with oXiris

INTERVENTIONS:
Device: Continuous renal replacement therapy with oXiris — Continuous renal replacement therapy with oXiris in patient with septic shock

SUMMARY:
The objectives of this study are to determine whether Continuous Renal Replacement Therapy (CRRT) with oXiris in patients with septic shock would improve clinical outcomes such as the sepsis-related organ failure assessment (SOFA) , hemodynamic, mortality compared CRRT with conventional membrane.

DETAILED DESCRIPTION:
Sepsis is the leading cause of death in ICU, resulting in multi-organ failure in critically ill patients. Patients with septic shock combined sepsis-associated Acute kidney injury (AKI)have even poorer outcome.

Endotoxin activity, inflammation and immune dysfunction, have been consider relevant to their pathogenesis of sepsis. High levels of Inflammation are associated with worse clinical outcomes. However, all studies of anti-inflammation treatment in sepsis patient are failed and anti-inflammation treatment of sepsis still remains controversial.

oXiris is a new filter with adsorptive membrane, which removes endotoxin and inflammatory mediator from plasma. But current evidence of oXiris is limited, and only some small sample studies have proved that it can improve the haemodynamics and the sepsis-related organ failure assessment(SOFA) score.

Our hypothesis was that oXiris would be associated with better clinical outcomes, such as decreased SOFA score, improved survival rate, better hemodynamic, and improved of organ function.

ELIGIBILITY:
Inclusion Criteria:

* >18 Years
* Treated by CRRT using oXiris or conventional membrane
* SOFA cardiovascular Score ≥ 3
* Septic shock due to abdominal or pneumonia( Gram-negative bacterial infection or suspected GNB infection)
* Written informed consent

Exclusion Criteria:

* Chronic Kidney Disease
* Renal replacement therapy (RRT) in the last 30 days
* Pregnancy
* Immunosuppressive treatment or steroids (prednisone > 0.5 mg/kg/day or equivalent).
* Autoimmune disorder.
* Transplant receptor.
* Inclusion in other ongoing studies within the last 30 days.
* Coexisting illness with a high probability of death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic shock patients due to abdominal or pneumonia( Gram-negative bacterial infection or suspected GNB infection) treated by CRRT
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  28-day mortality
The Sepsis-related Organ Failure Assessment(SOFA) cardiovascular Scores at 72 hours | 72 hours after Continuous Renal Replacement Therapy initiation
  The Sepsis-related Organ Failure Assessment(SOFA) cardiovascular Scores at 72 hours(Scores Range 0-4, higher values represent a worse outcome)

SECONDARY OUTCOMES:
Changes of Sepsis-related Organ Failure Assessment(SOFA) Score | 72 hours after Continuous Renal Replacement Therapy initiation
  Changes from baseline to 72 hours in Sepsis-related Organ Failure Assessment(SOFA) Score
VIS-Norepinephrine dose or equivalent | 72 hours after Continuous Renal Replacement Therapy initiation
  Norepinephrine dose or equivalent at 72 hours after Continuous Renal Replacement Therapy initiation
Change of Norepinephrine dose Over Time | 72 hours after Continuous Renal Replacement Therapy initiation
  Difference of Norepinephrine dose at 72 hours compared with Continuous Renal Replacement Therapy initiation
Vasopressor-free days | Day 28
  Vasopressor-free days to day 28
Lactate concentration at 72 hours | 72 hours after Continuous Renal Replacement Therapy initiation
  Lactate concentration level at 72 hours after Continuous Renal Replacement Therapy initiation initiation
ICU mortality | through study completion, an average of 1 month
  All cause mortality in ICU
mechanical ventilation free days | Day 28
  Total length of mechanical ventilation free days up to to day 28
Total length of Continuous Renal Replacement Therapy | Day 28
  Total length of Continuous Renal Replacement Therapy to day 28

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Department of Nephrology, Sichuan University West ChinaHospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make individual participant data (IPD) available to other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: The corresponding author will review requests form and provide the IPD

REFERENCES:
- [Background] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- [Background] Shum HP, Chan KC, Tam CW, Yan WW, Chan TM. Impact of renal replacement therapy on survival in patients with KDIGO stage 3 acute kidney injury: A propensity score matched analysis. Nephrology (Carlton). 2018 Dec;23(12):1081-1089. doi: 10.1111/nep.13164. PMID 28898482
- [Background] Peerapornratana S, Manrique-Caballero CL, Gomez H, Kellum JA. Acute kidney injury from sepsis: current concepts, epidemiology, pathophysiology, prevention and treatment. Kidney Int. 2019 Nov;96(5):1083-1099. doi: 10.1016/j.kint.2019.05.026. Epub 2019 Jun 7. PMID 31443997
- [Background] SepNet Critical Care Trials Group. Incidence of severe sepsis and septic shock in German intensive care units: the prospective, multicentre INSEP study. Intensive Care Med. 2016 Dec;42(12):1980-1989. doi: 10.1007/s00134-016-4504-3. Epub 2016 Sep 29. PMID 27686355
- [Background] Fani F, Regolisti G, Delsante M, Cantaluppi V, Castellano G, Gesualdo L, Villa G, Fiaccadori E. Recent advances in the pathogenetic mechanisms of sepsis-associated acute kidney injury. J Nephrol. 2018 Jun;31(3):351-359. doi: 10.1007/s40620-017-0452-4. Epub 2017 Dec 23. PMID 29273917
- [Background] Dellinger RP, Bagshaw SM, Antonelli M, Foster DM, Klein DJ, Marshall JC, Palevsky PM, Weisberg LS, Schorr CA, Trzeciak S, Walker PM; EUPHRATES Trial Investigators. Effect of Targeted Polymyxin B Hemoperfusion on 28-Day Mortality in Patients With Septic Shock and Elevated Endotoxin Level: The EUPHRATES Randomized Clinical Trial. JAMA. 2018 Oct 9;320(14):1455-1463. doi: 10.1001/jama.2018.14618. PMID 30304428
- [Background] Perez-Fernandez X, Sabater-Riera J, Sileanu FE, Vazquez-Reveron J, Ballus-Noguera J, Cardenas-Campos P, Betbese-Roig A, Kellum JA. Clinical variables associated with poor outcome from sepsis-associated acute kidney injury and the relationship with timing of initiation of renal replacement therapy. J Crit Care. 2017 Aug;40:154-160. doi: 10.1016/j.jcrc.2017.03.022. Epub 2017 Mar 30. PMID 28407544
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Result] Bouchard J, Acharya A, Cerda J, Maccariello ER, Madarasu RC, Tolwani AJ, Liang X, Fu P, Liu ZH, Mehta RL. A Prospective International Multicenter Study of AKI in the Intensive Care Unit. Clin J Am Soc Nephrol. 2015 Aug 7;10(8):1324-31. doi: 10.2215/CJN.04360514. Epub 2015 Jul 20. PMID 26195505